CLINICAL TRIAL: NCT00655200
Title: Observational Study of Safety and Tolerability of Levemir™ FlexPen™ (Insulin Detemir) in the Treatment of Type 1 and Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3525
Record Dates: First submitted 2008-04-04; First posted 2008-04-09 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Start dose and frequency to be prescribed by the physician as a result of the normal clinical evaluation
  Other Names: Levemir™

SUMMARY:
This study is conducted in Asia. The aim of this observational study is to evaluate the safety and tolerability of Levemir™ FlexPen™ (Insulin Detemir) in the treatment of Filipino patients with Type 1 and Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Type 1 or Type 2 Diabetes Mellitus.
* Newly diagnosed insulin naive patients
* Patients currently on human insulin or on basal insulin
* Patients prescribed with Levemir™ FlexPen™ (Insulin Detemir) therapy
* Usage should be in accordance with the current prescribing information (See attached prescribing information)

Exclusion Criteria:

* Previous history of hypersensitivity to Insulin Detemir (Levemir™) and its excipients (See attached prescribing information)
* Contraindications and warnings specified in the current prescribing information (See attached prescribing information)
* Pregnant women, those planning to become pregnant, or women who are breastfeeding
* Patients who are already on human premix or premix analogue (unless they are going to be shifted to basal-bolus therapy)
* Children below 6 years old

Ages: 0 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with Type 1 and Type 2 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 2286 (Actual)
Dates: Start 2008-02; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Safety profile of Insulin Detemir among Filipino patients | 3 months follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Manila, Philippines

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com